CLINICAL TRIAL: NCT04930198
Title: PeerNaija: A Mobile Health Platform Incentivizing Medication Adherence Among Youth Living With HIV in Nigeria
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); APIN Public Health Initiatives (Unknown); Nigerian Institute of Medical Research (Other Government); Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Martin C. Were, Professor Biomedical Informatics and Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 200116; R21TW011327 (NIH)
Record Dates: First submitted 2021-05-25; First posted 2021-06-18 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: HIV/AIDS
Keywords: HIV/AIDS; Sub-Saharan Africa
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Social Incentive (Other): For the social incentive, the mHealth application will track the participant's individual adherence score (% of doses taken), track the top scorers (leaderboard), and provide a figure highlighting the proportion of their peers with poor (<80%), medium (80-94%), or high (>94%) adherence scores. The display of the individual's adherence score relative to peer scores is considered a descriptive norm and is meant to portray "what most people are doing," as young people often inaccurately estimate behaviors for their peer groups. Participants will also receive an injunctive norm, or an indication of what they ought to be doing. This will come in the form of an emoji or congratulatory vs. motivating text for those with high or low adherence scores, respectively. When coupled with descriptive norms, injunctive norms have counteracted regression to the mean for individuals who demonstrate desirable behaviors relative to their peers.
  Interventions: Behavioral: PeerNaija
- Social Plus Financial Incentive (Other): For the financial incentive, the top 5 scorers in the PEER+ arm will be eligible win a lottery prize each month of the 24 week pilot of 1000 Nigerian Naira (NGN) of "data" that can be directly loaded onto the winner's phone. Behavioral economics theory tells us that individuals are more averse to losses than rewarded by gains, so that even incentives/prizes should be framed in terms of losses. Accordingly, participants in the financial incentive arm will receive weekly motivating messages such as "take your dose today or you lose the chance of winning the lottery."
  Interventions: Behavioral: PeerNaija

INTERVENTIONS:
Behavioral: PeerNaija — All participants (anticipated N=50) will receive daily medication reminders and access to the virtual support group on the PEERNaija app. Participants will be randomized to receive a social incentive (anticipated n=25) or a social plus financial incentive (anticipated n=25), PEER+, and be followed for 24 weeks.

SUMMARY:
The PEERNaija application will feature routine medication reminders, along with individual adherence monitoring with adherence scores, anonymized peer adherence scores (from peers attending the same clinic; social incentive), and a monthly lottery-based prize for youth with the highest adherence scores (financial incentive). The Investigators will recruit a cohort of 50 HIV-infected adolescents and young adults (AYA) to pilot the app and assess feasibility, acceptability, adoption, and preliminary efficacy of important clinical measures (including adherence and virologic suppression). The proposed study will provide important preliminary data for the role of mobile health (mHealth) platforms to harness and deliver social and financial incentives to promote adherence efforts, especially for vulnerable youth, and for a larger intervention trial evaluating this app among HIV-infected AYA in Nigeria.

DETAILED DESCRIPTION:
The use of digital health solutions, especially medication reminders delivered via mHealth platforms, have shown promise as adherence support tools in sub-Saharan Africa (SSA). Importantly, the proliferation of mobile phones in resource-limited settings and the early adoption of communication technologies by young people make mHealth technologies an ideal platform for this age group. The Investigators propose to pilot a novel, mHealth peer-based intervention for AYA living with HIV in Nigeria that will utilize social and financial incentives to promote medication adherence. In addition to medication reminders and peer support, the proposed intervention will innovate within the mHealth arena to leverage the currency of social incentives through daily adherence monitoring with the provision of adherence scores for individual users in relation to their peers, and financial incentives through a monthly lottery for youth with the highest adherence scores with the prize delivered through the mHealth application itself. This proposal builds on the Investigator's successful research collaborations in Nigeria with APIN Public Health Initiatives, (APIN, a multi-site non-governmental organization with solid President's Emergency Plan For AIDS Relief-funded HIV infrastructure), the investigators expertise in building capacity for implementation research, and proficiency in developing and deploying mHealth-based interventions in SSA. This will be accomplished through the following specific aim:

To establish the feasibility, acceptability, and preliminary efficacy of PEERNaija, an mHealth intervention designed to harness peer influence as an incentive to promote medication adherence among a pilot cohort of 50 AYA living with HIV in Nigeria. Hypothesis: PEERNaija will be feasible, acceptable, and show preliminary efficacy in improving antiretroviral (ART) adherence.

ELIGIBILITY:
Inclusion Criteria:

* Own a smartphone (on which they are willing to download PEERNaija),
* 16-27 years of age,
* on ART, and
* demonstrate the ability read simple text language in English.

Ages: 16 Years to 27 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aima Ahonkhai, MD, MPH, Principal Investigator — Massachusetts General Hospital; Martin C Were, MD, MS, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- Nigeria (2):
  - APIN Public Health Initiatives, Abuja
  - Nigerian Institute of Medical Researd, Lagos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Were MC, Pierce LJ, Idigbe I, Okonkwo P, Mbugua S, Savai S, Eliazer CL, Ahonkhai AA. Applying Gamification Principles to a Mhealth App to Support Adherence to Hiv Medication in a Resource-Limited Setting. Stud Health Technol Inform. 2025 Aug 7;329:1545-1549. doi: 10.3233/SHTI251098. PMID 40776116
- [Result] Idigbe I, Were M, Pierce LJ, Ekelem C, Nmoh A, Gbaja-Biamila T, David A, Ejiga Q, Ogunwale J, Adetoye D, Okonkwo P, Musa Z, Downshen N, Ezechi O, Audet C, Ahonkhai AA. User-centered adaption of PEERNaija, A novel mhealth application integrating medication reminders with virtual peer support and social/financial incentives to improve medication adherence. AIDS Care. 2025 Feb;37(2):263-278. doi: 10.1080/09540121.2024.2445789. Epub 2025 Jan 6. PMID 39761419
- [Result] Ahonkhai AA, Pierce LJ, Mbugua S, Wasula B, Owino S, Nmoh A, Idigbe I, Ezechi O, Amaral S, David A, Okonkwo P, Dowshen N, Were MC. PEERNaija: A Gamified mHealth Behavioral Intervention to Improve Adherence to Antiretroviral Treatment Among Adolescents and Young Adults in Nigeria. Front Reprod Health. 2021;3:656507. doi: 10.3389/frph.2021.656507. Epub 2021 Jul 30. PMID 35237765
- [Result] Pierce LJ, Were MC, Amaral S, Aliyu MH, Ezechi O, David A, Idigbe I, Musa AZ, Okonkwo P, Dowshen N, Ahonkhai AA. PEERNaija-a mobile health platform incentivizing medication adherence among youth living with HIV in Nigeria: study protocol for a randomized controlled trial. Pilot Feasibility Stud. 2023 Oct 27;9(1):179. doi: 10.1186/s40814-023-01404-0. PMID 37891681

RESULTS

PARTICIPANT FLOW:
Groups:
- Social Incentive: For the social incentive, the mHealth application will track the participant's individual adherence score (% of doses taken), track the top scorers (leaderboard), and provide a figure highlighting the proportion of their peers with poor (<80%), medium (80-94%), or high (>94%) adherence scores. The display of the individual's adherence score relative to peer scores is considered a descriptive norm and is meant to portray "what most people are doing," as young people often inaccurately estimate behaviors for their peer groups. Participants will also receive an injunctive norm, or an indication of what they ought to be doing. This will come in the form of an emoji or congratulatory vs. motivating text for those with high or low adherence scores, respectively. When coupled with descriptive norms, injunctive norms have counteracted regression to the mean for individuals who demonstrate desirable behaviors relative to their peers.
  PeerNaija: All participants (N=50) will receive daily medication reminders and access to the virtual support group on the PEERNaija app. Participants will be randomized to receive a social incentive (n=25) or a social plus financial incentive (n=25), PEER+, and be followed for 24 weeks.
- Social Plus Financial Incentive: For the financial incentive, the top 5 scorers in the PEER+ arm will be eligible win a lottery prize each month of the 24 week pilot of 1000 Nigerian Naira (NGN) of "data" that can be directly loaded onto the winner's phone. Behavioral economics theory tells us that individuals are more averse to losses than rewarded by gains, so that even incentives/prizes should be framed in terms of losses. Accordingly, participants in the financial incentive arm will receive weekly motivating messages such as "take your dose today or you lose the chance of winning the lottery."
  PeerNaija: All participants (N=50) will receive daily medication reminders and access to the virtual support group on the PEERNaija app. Participants will be randomized to receive a social incentive (n=25) or a social plus financial incentive (n=25), PEER+, and be followed for 24 weeks.
Period: Overall Study
Arm/Group | Social Incentive | Social Plus Financial Incentive
Started | 26 | 28
Completed | 19 | 23
Not Completed | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Social Incentive | Social Plus Financial Incentive | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.3 (2.8) | 19.2 (3.9) | 18.8 (3.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 14 | 13 | 27
  Female | 10 | 14 | 24
  Unknown | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 28 | 54
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Nigeria | 26 | 28 | 54
Baseline Viral Load [Mean (Standard Deviation); unit: copies/mL] | 14327.1 (41822.3) | 6010.2 (27266.1) | 9422.3 (33734.7)

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: Recruitment rate is measured by the percentage of participants randomized relative to total trial referrals.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Groups:
- Social Incentive: For the social incentive, the mHealth application will track the participant's individual adherence score (% of doses taken), track the top scorers (leaderboard), and provide a figure highlighting the proportion of their peers with poor (<80%), medium (80-94%), or high (>94%) adherence scores. The display of the individual's adherence score relative to peer scores is considered a descriptive norm and is meant to portray "what most people are doing," as young people often inaccurately estimate behaviors for their peer groups. Participants will also receive an injunctive norm, or an indication of what they ought to be doing. This will come in the form of an emoji or congratulatory vs. motivating text for those with high or low adherence scores, respectively. When coupled with descriptive norms, injunctive norms have counteracted regression to the mean for individuals who demonstrate desirable behaviors relative to their peers.
  PeerNaija: All participants (anticipated, N=50) will receive daily medication reminders and access to the virtual support group on the PEERNaija app. Participants will be randomized to receive a social incentive (anticipated, n=25) or a social plus financial incentive (anticipated, n=25), PEER+, and be followed for 24 weeks.
- Social Plus Financial Incentive: For the financial incentive, the top 5 scorers in the PEER+ arm will be eligible win a lottery prize each month of the 24 week pilot of 1000 Nigerian Naira (NGN) of "data" that can be directly loaded onto the winner's phone. Behavioral economics theory tells us that individuals are more averse to losses than rewarded by gains, so that even incentives/prizes should be framed in terms of losses. Accordingly, participants in the financial incentive arm will receive weekly motivating messages such as "take your dose today or you lose the chance of winning the lottery."
  PeerNaija: All participants (anticipated, N=50) will receive daily medication reminders and access to the virtual support group on the PEERNaija app. Participants will be randomized to receive a social incentive (anticipated, n=25) or a social plus financial incentive (anticipated, n=25), PEER+, and be followed for 24 weeks.
Arm/Group | Social Incentive | Social Plus Financial Incentive
Number analyzed (Participants) | 26 | 28
Participants | 26 | 28

2. Primary Outcome: Retention Rate
Description: Retention rate is measured by the percentage of participants who completed the 24-week follow-up.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Social Incentive | Social Plus Financial Incentive
Number analyzed (Participants) | 26 | 28
Participants | 19 | 23

3. Primary Outcome: Feasibility of Intervention
Description: Feasibility will be assessed with the Feasibility of Intervention Measure (FIM), a validated, four-item measure to determine the extent to which stakeholders believe an intervention is feasible to implement. The FIM will assess participant's likes/dislikes of the mobile health platform, privacy/security concerns, technology barriers, usage preferences, medication compliance and reasons for non-compliance. The FIM is scored on a scale of 1-5 with higher scores indicating higher perceived feasibility.
Time Frame: 24 weeks
Population: FIM is a validated tool; if a participant skipped any single item, their score was counted as missing and they were excluded from data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Incentive | Social Plus Financial Incentive
Number analyzed (Participants) | 18 | 22
score on a scale | 4.0 (0.7) | 4.0 (0.7)

4. Primary Outcome: Acceptability of Intervention
Description: Acceptability will be assessed with the Acceptability of Intervention Measure (AIM), a validated, four-item measure to determine the extent to which stakeholders believe an intervention is feasible to implement. The AIM will assess participant's likes/dislikes of the mobile health platform, privacy/security concerns, technology barriers, usage preferences, medication compliance and reasons for non-compliance. The AIM is scored on a scale of 1-5 with higher scores indicating higher perceived acceptability.
Time Frame: 24 weeks
Population: AIM is a validated tool; if a participant skipped any single item, their score was counted as missing and they were excluded from data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Incentive | Social Plus Financial Incentive
Number analyzed (Participants) | 18 | 22
score on a scale | 4.2 (0.6) | 4.0 (0.7)

5. Primary Outcome: Appropriateness of Intervention
Description: Appropriateness will be assessed with the Intervention Appropriateness Measure (IAM), a validated, four-item measure to determine the extent to which stakeholders believe an intervention is feasible to implement. The IAM will assess participant's likes/dislikes of the mobile health platform, privacy/security concerns, technology barriers, usage preferences, medication compliance and reasons for non-compliance.
Time Frame: 24 weeks
Population: The IAM is scored on a scale of 1-5 with higher scores indicating higher perceived appropriateness. IAM is a validated tool; if a participant skipped any single item, their score was counted as missing and they were excluded from data analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Social Incentive | Social Plus Financial Incentive
Number analyzed (Participants) | 18 | 22
score on a scale | 4.2 (0.6) | 4.0 (0.8)

6. Primary Outcome: Preliminary Efficacy of Intervention on Viral Load
Description: Preliminary efficacy will be assessed by identifying the number of participants virally suppressed at study end (undetectable < 1000 m/ml).
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Social Incentive | Social Plus Financial Incentive
Number analyzed (Participants) | 19 | 23
Participants | 16 | 18

ADVERSE EVENTS:
Time Frame: 6 months.
Description: All serious and non-serious adverse events were collected systematically during the study period in line with the study's data collection plan. The study's definitions of adverse event and/or serious adverse event were as defined in clinicaltrials.gov.
Groups:
- Social Incentive: No breaches in confidentiality or other attributable adverse events occurred in the 'Social Incentive' group over the study period.
- Social Plus Financial Incentive: No breaches in confidentiality or other attributable adverse events occurred to the 'Social Plus Financial Incentive' over the study period.
Arm/Group | Social Incentive | Social Plus Financial Incentive
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/28
Other Adverse Events (participants affected / at risk) | 0/26 | 0/28

LIMITATIONS AND CAVEATS:
As a pilot, the trial recruited a small sample size. Otherwise, we have nothing to report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-10-05): https://cdn.clinicaltrials.gov/large-docs/98/NCT04930198/Prot_SAP_001.pdf
  • Informed Consent Form (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT04930198/ICF_000.pdf